Title: Physical Literacy-based Intervention (PLBI) for Older Adults: A Cluster Randomized Controlled Trial Study Protocol

NCT number: NCT06137859

**Date of document: 24/08/2024** 



## The Chinese University of Hong Kong

### **Consent Form**

Project title: Physical literacy-based intervention (PLBI) for older adults: a cluster

randomized controlled trial

Investigator: Sum Kim Wai, Raymond

Department of Sports Science & Physical Education (SSPE)

The Chinese University of Hong Kong (CUHK)

First of all, thank you for your interest to take part in this project. Please take your time to review this consent form and discuss any questions you may have, or words you do not clearly understand, with the investigator or staff.

#### **Purpose of the Study**

The purpose of this study is to explore physical literacy (physical competency, daily behavior, knowledge and understanding, and motivation and confidence) of the older adults in Hong Kong

## **Voluntary Participation**

Your participation is completely voluntary and you may withdraw your participation at any time during the process, either temporarily or permanently.

#### **Study Procedures**

Upon receiving your consent, you will be contacted by phone and, or, email according to your preferred contact. In this project, should you decide to participate, you will be allocated into one of the two groups - intervention and control group. You will be notified by e-mail and telephone about their randomization allocation. Before and after a twelve-week intervention, you will be requested to complete questionnaires of physical literacy, motivation and confidence and PA engagement, together with a cognitive test and objective physical competence assessment. These measurements will be completed again by all of the participants six weeks after the intervention period.

Your participation will be able to contribute valuable insights to the conceptual framework of developing physical literacy program for older adults in Hong Kong. And in the long run, due to the feasibility and sustainability of these potential programs, this proposed project has the potential to connect seniors through social engagement and contribute to intergenerational-healthy-living.

# **Confidentiality**

Your participation in this study will be strictly confidential. Your real name will not be used at the intervention. No identifying information and name will be used and revealed in any written reports or publications. All findings in this study will be reported in aggregate form with no identifying information.

| Should any questions arise at any point during the study, please do not hesitate to contact me at: 3943 6091 (office), or 9217 4388 (mobile). | | |
|---|---|---|
| Signature of Investigator | Date | |
| Info | mant's Consent | |
| • | ritten consent to the study discussed above. I als all the relevant materials with regards to my ant queries have been responded to my | O |
| Signature of Investigator | Date | |